CLINICAL TRIAL: NCT01832532
Title: Pilot 2: Glucagon-like Peptide-1 in Sleep Disordered Breathing
Brief Title: A Pilot Study of the Effects on Sleep Disordered Breathing (SDB) When Using the Drug Liraglutide for 4 Weeks
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIN001Pilot 2GLP; UL1RR026314 (NIH)
Record Dates: First submitted 2013-04-08; First posted 2013-04-16 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Sleep Apnea; Sleep Disordered Breathing
Keywords: Sleep Apnea; Sleep Disordered Breathing; liraglutide; glucagon-like peptide-1 agonist; Orexin; leptin,
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group- liraglutide (Experimental): Treatment group- liraglutide daily use of drug. Titrated up from 0.6mg/day to 1.8mg/day or highest tolerated dose.
  Interventions: Drug: liraglutide
- Control group (No Intervention): Control group

INTERVENTIONS:
Drug: liraglutide — daily use of drug. Titrated up from 0.6mg/day to 1.8mg/day or highest tolerated dose
  Other Names: Other name- Victoza
  Arms: Treatment group- liraglutide

SUMMARY:
This is an open label, controlled study.

The investigators are studying if the FDA approved diabetes medicine liraglutide (Victoza®) can improve sleep apnea in adults. This study is testing liraglutide in 20 adults without diabetes that are diagnosed with sleep apnea.The treatment group will be compared to a control group of 10 adults without diabetes who have sleep apnea but will not use liraglutide. Both groups will continue receiving standard of care for their sleep apnea as prescribed by their managing sleep physician throughout their study participation.

Everyone in the study will have two study visits and one overnight sleep study for research. Subjects who have not had a recent sleep study but otherwise qualify for the study, will have an additional research sleep study to determine the baseline severity of their sleep apnea. The study visits include fasting blood samples and breathing tests (pulmonary function test and hypercapnic challenge). There will be weekly phone visits that include a questionnaire on sleepiness. The group that takes liraglutide will check their blood sugar two times a day while on the medicine.

DETAILED DESCRIPTION:
This is a pilot study aimed at measuring the change in obstructive apnea/hypopnea index in non-diabetic patients being treated for the first time with the glucagon-like peptide-1 (GLP-1) agonist, Liraglutide. Sleep disordered breathing (SDB) consists of nocturnal alveolar hypoventilation and / or obstructive sleep apnea which result from abnormalities in upper airway tone and ventilation during sleep. The development of a new pharmacological treatment for sleep disordered breathing (SDB) could bring a breakthrough discovery that will impact a rapidly growing population of children and adults with this disorder. The investigators hypothesize that GLP-1 plays a central role in the improvement of SDB and that the administration of GLP-1 receptor agonist to patients with OSA will correct or improve SDB.

* Hypothesis 1: Administration of Liraglutide to patients with severe OSA defined as apnea hypopnea index ≥ 8 /hr. will result in a mean reduction in the index by a minimum of 50% after 4 weeks.
* Hypothesis 2: Administration of Liraglutide will result in significant increase in Orexin level, decrease in leptin, decrease in Epworth Sleepiness Scale (ESS) score and increase in carbon dioxide (CO2) chemosensitivity.

This is an open label, non-randomized, controlled pilot study. Subjects are heavy to obese non-diabetic adults that are diagnosed with sleep apnea. 20 subjects will be treated with liraglutide for 4 weeks and compared to 10 untreated controls.

Study time points are baseline and 4 weeks post treatment. Study procedures include pre and post treatment: fasting blood for glucose, hemoglobin A1C (HbA1C), Orexin and leptin; ESS questionnaire; pulmonary function test and hypercapnic challenge. The procedures also include a post treatment overnight research sleep study to measure change in apnea index from diagnostic sleep study done previous to study enrollment or if needed, the baseline research sleep study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Diagnosis of severe obstructive sleep apnea (OSA) AHI ≥ 8 /hour of sleep
* Ability and willingness to comply with all protocol procedures e.g. correct handling of trial product, compliance to visit schedule
* BMI of ≥ 27
* For Cohort 1: If female of childbearing capacity, willing to use acceptable birth control during use of study drug

Exclusion Criteria:

* A major medical condition such as renal or hepatic failure
* Treatment with glucagon-like peptide-1 (GLP-1) receptor agonists, dipeptidyl peptidase-4 inhibitors or insulin within the last 3 months prior to screening
* Diagnosis of type 1 or type 2 diabetes per judgment of the investigator
* BMI < 27
* History of glycosylated hemoglobin (HbA1c) equal to or above 6.5%
* Significant craniofacial abnormalities that may cause OSA
* Respiratory and neuromuscular diseases that could interfere with the results of the trial in the opinion of the investigator
* Use of central stimulants, hypnotics, mirtazepine, opioids, trazodone or drugs in the incretin family within the previous 3 months prior to screening
* Previous surgical treatment for obesity
* Familial or personal history of Multiple Endocrine Neoplasia type 2 or familial Medullary Thyroid Carcinoma
* Personal or immediate family history of thyroid cancer
* History of chronic pancreatitis or idiopathic acute pancreatitis
* History of Major Depressive Disorder or suicide attempts
* Systolic blood pressure equal to or above 160 mmHg and/or diastolic blood pressure equal to or above 100 mmHg
* History of alcoholism
* Pregnancy or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raouf Amin, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Manuscript is in progress.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment fell short of goal for each cohort
Period: Overall Study
Arm/Group | Treatment Group- Liraglutide | Control Group
Started | 23 | 11
Completed | 18 | 9
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group- Liraglutide | Control Group | Total
Number analyzed (Participants) | 18 | 9 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 9 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (8) | 44.5 (10.6) | 46.2 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 13 | 7 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 16 | 7 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Apnea Hypopnea Index (AHI) From Baseline
Description: Change in the number of apneas plus hypopnea events per hour of sleep from baseline at end of study.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: apnea / hypopnea events per hour sleep
Arm/Group | Treatment Group- Liraglutide | Control Group
Number analyzed (Participants) | 18 | 9
apnea / hypopnea events per hour sleep | 38.2 (30) | 34 (20)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Treatment Group- Liraglutide | Control Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/9
Other Adverse Events (participants affected / at risk) | 0/18 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No